CLINICAL TRIAL: NCT03251261
Title: Illumigene CMV Clinical Trial Protocol
Brief Title: Detection of Cytomegalovirus Virus in Neonates
Acronym: CMV
Status: Completed | Type: Observational
Sponsor: Meridian Bioscience, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CLIN-DHF-333-001
Record Dates: First submitted 2017-08-14; First posted 2017-08-16 (Actual); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: CMV

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Prospectively collected saliva swabs from neonates up to 21 days of age Retrospective well characterized positive saliva samples will also be tested
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Specimen collection
  Interventions: Device: illumigene CMV assay, illumipro-10

INTERVENTIONS:
Device: illumigene CMV assay, illumipro-10 — CMV assay for detection of CMV

SUMMARY:
To evaluate the illumigene CMV assay, using the illumipro-10 with neonates (up to 21 days of age) saliva swabs

ELIGIBILITY:
Inclusion Criteria:

* Saliva swab specimens from neonates up to 21 days of age
* Saliva swab sample placed in a nonnutritive transport medium or in a plastic sterile tube without medium.
* Flocked-nylon swabs

Exclusion Criteria:

* Samples other than saliva swab from patients up to 21 days of age.
* Swabs other than flocked-nylon.
* Swabs in a viral transport media not defined in the Investigational Use Only package insert
* Multiple specimens from the same patient.
* Specimens received in the laboratory in unsatisfactory containers or condition.

Max Age: 20 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Saliva swab specimens from all neonates up to 21 days of age may be collected and tested
Sampling Method: Non-Probability Sample
Enrollment: 1615 (Actual)
Dates: Start 2017-08-02 (Actual); Primary Completion 2018-03-05 (Actual); Study Completion 2018-03-05 (Actual)

PRIMARY OUTCOMES:
Qualitative detection of CMV to aid in the diagnosis of CMV | within 30 days of sample collection
  Test each sample for CMV detection

CONTACTS AND LOCATIONS:
Overall Officials: Julie M Kesler, Study Director — Meridian Bioscience; Ken Kozak, Study Chair — Meridian Bioscience
Locations (5):
- United States (2):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Utah, Salt Lake City, Utah
- The Prince of Wales Hospital, Randwick, New South Wales, Australia
- British Columbia Children's Hospital / British Columbia Women's Hospital, Vancouver, British Coloumbia, Canada
- Ospedale Sant'Orsola, Via Massarenti 19, Province of Bologna, Italy